CLINICAL TRIAL: NCT01835054
Title: Determinants of the Progression and Outcome of Mitral Regurgitation-PROGRAM STUDY
Brief Title: Determinants of the Progression and Outcome of Mitral Regurgitation
Acronym: PROGRAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other); University Hospital, Brest (Other)
Responsible Party: Principal Investigator, Philippe Pibarot, Doctor, Laval University
Other Study IDs: MOP#102737
Record Dates: First submitted 2013-04-16; First posted 2013-04-18 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Mitral Valve Insufficiency
Keywords: Mitral regurgitation; Mitral valve prolapse; Echocardiography, Doppler; Stress echocardiography; Cardiopulmonary exercice testing; Magnetic Resonance Imaging; Cardiac neurohormones; Visceral obesity; Cardiometabolic risk; Risk stratification
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Obesity, Abdominal | interventions — Exercise Test; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fasting blood sample (serum, lithium-heparin, EDTA) and white cells - Tissue (explanted mitral valves)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with mitral regurgitation: At study entry, patients have 1) a clinical assessment including metabolic risk profile; 2) a blood sample for analysis of metabolic, cardiac neurohormonal blood biomarkers and DNA collection; 3) a complete rest doppler echocardiography; 4) an exercise stress doppler echocardiography; 5) a cardiopulmonary exercise testing; 6) a magnetic resonance Imaging (MRI); 7) a 24-hour Holter ECG.
  At follow-up, patients have 1) a clinical events assessment; 2) a blood sample analysis; 3) a resting echocardiography every year; 4) MRI (at preop. evaluation in the subset of patients undergoing surgery); 5) a 24-hour Holter ECG (at 2-year and postop.).
  Interventions: Other: Blood biomarkers; Genetic: DNA collection; Other: Echocardiography; Other: Cardiopulmonary exercise testing; Other: Magnetic resonance imaging (MRI); Other: Exercise stress doppler echocardiography; Other: Holter ECG

INTERVENTIONS:
Other: Blood biomarkers — Observational Study using Imaging and Biomarkers
Genetic: DNA collection — Observational Study using Imaging and Biomarkers
Other: Echocardiography — Observational Study using Imaging and Biomarkers
Other: Cardiopulmonary exercise testing — Observational Study using Imaging and Biomarkers
Other: Magnetic resonance imaging (MRI) — Observational Study using Imaging and Biomarkers
Other: Exercise stress doppler echocardiography — Observational Study using Imaging and Biomarkers
Other: Holter ECG — Observational Study using Imaging and Biomarkers

SUMMARY:
Mitral regurgitation (MR) is one of the most frequent valve lesions, both in North America and in Europe, and its prevalence is increasing with the aging of the population. Organic Mitral Regurgitation (OMR) and Ischemic Mitral Regurgitation are the 2 main categories of MR. Organic or primary MR is caused by an anatomic alteration of the valvular or subvalvular mitral apparatus and refers to rheumatic MR and degenerative MR that includes mitral leaflet prolapse and flail leaflet. In the past 20 years, degenerative MR has become, by far, the most frequent cause of severe MR leading to surgery in the western world. However, the best current treatment for OMR remains uncertain and controversial. We have obtained preliminary data showing that OMR is a dynamic lesion. Hence, the echocardiographic evaluation of MR at rest, as generally performed during routine clinical exam, does not necessarily reflect the status of MR during patient's daily activities and thereby does not adequately assess the risk of rapid progression and poor outcome in these patients. The objective of this study is to identify the independent predictors of disease progression and outcome in patients with asymptomatic chronic OMR and to develop and validate novel imaging and circulating biomarkers to improve risk stratification and therapeutic decision-making process in patients with chronic asymptomatic primary OMR.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) is one of the most frequent valve lesions, both in North America and in Europe, and its prevalence is increasing owing to the aging of the population. There are 2 main categories of MR: Organic Mitral Regurgitation (OMR) and Ischemic Mitral Regurgitation. Organic or primary MR is caused by an anatomic alteration of the valvular or subvalvular mitral apparatus and refers to rheumatic MR and degenerative MR that includes mitral leaflet prolapse and flail leaflet. In the past 20 years, degenerative MR has become, by far, the most frequent cause of severe MR leading to surgery in the western world. However, the best current treatment for OMR remains uncertain and controversial. This is, in large part, due to the lack of prospective data on the determinants of OMR progression and outcome. Furthermore, we have obtained preliminary data showing that OMR is a dynamic lesion. Hence, the echocardiographic evaluation of MR at rest, as generally performed during routine clinical exam, does not necessarily reflect the status of MR during patient's daily activities and thereby does not adequately assess the risk of rapid progression and poor outcome in these patients.

The general objective of this study is thus: to identify the independent predictors of disease progression and outcome in patients with asymptomatic chronic OMR and to develop and validate novel imaging and circulating biomarkers to improve risk stratification and therapeutic decision-making process in patients with chronic asymptomatic primary OMR.

The specific aims of the study are: (1) To obtain and analyze: a) the dynamic changes in MR severity, pulmonary arterial pressure, and LV function during exercise; b) the maximum exercise capacity; c) the metabolic profile; d) the plasma natriuretic peptides, e) the degree and localization of myocardial fibrosis measured by cardiac magnetic resonance Imaging (MRI); f) the blood markers of myocardial extracellular matrix (ECM) turnover; g) the progression of MR severity and LV dysfunction during follow-up; and h) the occurrence of adverse clinical outcomes (i.e. symptoms, LV dysfunction, atrial fibrillation (Holter ECG), pulmonary hypertension, heart failure, cardiovascular death) during follow-up in a series of 440 patients with at least moderate OMR and no symptoms at baseline. (2) To analyze the valve tissue samples explanted from the patients who will undergo mitral valve repair with quadrangular resection during follow-up in order to document the presence of lipids, inflammation, and expression of metalloproteinases (MMPs). (3) To obtain and analyze the postoperative changes in LV geometry and function, pulmonary arterial pressure, symptoms, and exercise capacity in the subset of patients who will undergo mitral valve surgery during follow-up. (4) To evaluate the usefulness of the exercise induced changes in MR severity, pulmonary arterial pressure, and LV function (i.e. contractile reserve), and of the blood levels of natriuretic peptides and ECM biomarkers for the prediction of rapid progression to LV dysfunction and adverse events. (5) To examine the relationship between the metabolic abnormalities linked to visceral obesity and the progression and outcome of OMR. (6) To determine, among the baseline clinical, echocardiographic, MRI, metabolic, and biomarkers variables, those which are independently associated with the progression of MR severity and LV dysfunction, and the occurrence of adverse clinical outcomes in patients with OMR.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 or 21 years (Legal age according to the countries involved in this study)
* Presence of at least mild chronic OMR defined as an ERO ≥10mm2 and/or a regurgitant volume ≥20mL

Exclusion Criteria:

* MR due to ischemic heart disease or cardiomyopathy
* > mild mitral stenosis, aortic regurgitation, aortic stenosis or pulmonary stenosis
* previous valve operation
* history of myocardial infarction or angiographycally documented coronary stenosis
* congenital or pericardial heart disease
* endocarditis
* contra-indication or inability to exercise
* pregnancy
* Class I or IIa indication for mitral valve operation according to the 2014 ACC/AHA/ESC guidelines
* Typical contraindications to contrast-enhanced MRI (surgery in the last 3 months, defibrillator, pericardial electrodes, brain surgery, aneurysm clipping, neurostimulator, electric stimulation device or magnetically activated, cochlear implant, insulin pump or medication delivery device, Swan-Ganz catheter)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort will be selected at primary care clinic
Sampling Method: Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2008-12; Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Combined clinical and echocardiographic endpoint | Patients will be followed for 10 years
  The primary outcome is the time to occurrence of the first composite end-point: development of symptoms, left ventricular (LV) dysfunction (LV Ejection Fraction<60% and/or LV end diastolic diameter >40mm), ventricular arrhytmia requiring hospitalization, mediaction and/or implantation of defibrillator, atrial fibrillation or flutter, pulmonary arterial hypertension (resting systolic pressure >50mmHg), occurence of pulmonary oedema, congestive heart failure or cardiovascular death.

SECONDARY OUTCOMES:
Progression of MR severity | Patients will be followed for 10 years
  The annualized progression rate of MR severity will be calculated as the difference between effective regurgitant orifice, regurgitant volume, and vena contracta width measured at baseline and those measured at the last follow-up divided by the time between the first and last examinations.
Progression of pulmonary arterial hypertension | Patients will be folowed for 10 years
  The annualized progression rate of resting systolic pulmonary arterial pressure will be calculated.
Progression of LV dysfuntion prior to surgery | Patients will be followed for 10 years
  The annualized progression rate of LVEF, LV end-systolic dimension, and LV myocardial global peak systolic velocities and global longitudinal strain will be calculated.
Maximum exercise capacity at baselin and following mitral valve surgery | Patients will be followed for 10 years
  Maximum exercise capacity at baseline as measured by the percentage of age and gender predicted VO2max. We will determine which are, among the clinical and Doppler-echocardiographic variables, the independent determinants of maximum exercise capacity at baseline. The baseline exercise capacity will also be used as an independent variable, i.e. we will determine if it is an independent predictor of the primary end-point and of the other secondary end-points
Composite end-point prior to mitral valve surgery | Patients will be followed for 10 years
  i.e. follow-up censored at surgery
Composite primary end-point after mitral vale surgery | Patients will be followed for 10 years
  i.e. time zero set at surgery
Mitral valve surgery | Patients will be followed for 10 years
  Motivated by the occurrence of symptoms, LV systolic dysfunction, atrial fibrillation, and/or resting pulmonary pressure > 50 mmHg.
Arrhythmic burden | Patients will be followed for 10 years
  Number and percentage of ventricular ectopic per 24 h, percent time in atrial fibrillation, or flutter per 24 h.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Pibarot, PhD, DVM, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (4):
- University Hospital of Sart Tilman, Liège, Belgium
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Canada
- France (2):
  - University Hospital (CHU) of Brest, Hôpital La Cavale Blanche, Brest
  - University Hospital of Rennes, Rennes

REFERENCES:
- [Background] Magne J, Mahjoub H, Pibarot P, Pirlet C, Pierard LA, Lancellotti P. Prognostic importance of exercise brain natriuretic peptide in asymptomatic degenerative mitral regurgitation. Eur J Heart Fail. 2012 Nov;14(11):1293-302. doi: 10.1093/eurjhf/hfs114. Epub 2012 Jul 10. PMID 22782970
- [Background] Magne J, Mahjoub H, Pierard LA, O'Connor K, Pirlet C, Pibarot P, Lancellotti P. Prognostic importance of brain natriuretic peptide and left ventricular longitudinal function in asymptomatic degenerative mitral regurgitation. Heart. 2012 Apr;98(7):584-91. doi: 10.1136/heartjnl-2011-301128. Epub 2012 Feb 18. PMID 22342982
- [Background] Lancellotti P, Magne J. Stress testing for the evaluation of patients with mitral regurgitation. Curr Opin Cardiol. 2012 Sep;27(5):492-8. doi: 10.1097/HCO.0b013e3283565c3b. PMID 22872130
- [Background] Senechal M, Michaud N, Machaalany J, Bernier M, Dubois M, Magne J, Couture C, Mathieu P, Bertrand OF, Voisine P. Relation of mitral valve morphology and motion to mitral regurgitation severity in patients with mitral valve prolapse. Cardiovasc Ultrasound. 2012 Jan 27;10:3. doi: 10.1186/1476-7120-10-3. PMID 22284298
- [Background] Van de Heyning CM, Magne J, Vrints CJ, Pierard L, Lancellotti P. The role of multi-imaging modality in primary mitral regurgitation. Eur Heart J Cardiovasc Imaging. 2012 Feb;13(2):139-51. doi: 10.1093/ejechocard/jer257. Epub 2011 Nov 29. PMID 22127625
- [Background] Magne J, Lancellotti P, O'Connor K, Van de Heyning CM, Szymanski C, Pierard LA. Prediction of exercise pulmonary hypertension in asymptomatic degenerative mitral regurgitation. J Am Soc Echocardiogr. 2011 Sep;24(9):1004-12. doi: 10.1016/j.echo.2011.04.003. Epub 2011 May 17. PMID 21592726
- [Background] Magne J, Lancellotti P, Pierard LA. Exercise-induced changes in degenerative mitral regurgitation. J Am Coll Cardiol. 2010 Jul 20;56(4):300-9. doi: 10.1016/j.jacc.2009.12.073. PMID 20633822
- [Background] Magne J, Lancellotti P, Pierard LA. Exercise pulmonary hypertension in asymptomatic degenerative mitral regurgitation. Circulation. 2010 Jul 6;122(1):33-41. doi: 10.1161/CIRCULATIONAHA.110.938241. Epub 2010 Jun 21. PMID 20566950
- [Background] Magne J, Mathieu P, Dumesnil JG, Tanne D, Dagenais F, Doyle D, Pibarot P. Impact of prosthesis-patient mismatch on survival after mitral valve replacement. Circulation. 2007 Mar 20;115(11):1417-25. doi: 10.1161/CIRCULATIONAHA.106.631549. Epub 2007 Mar 5. PMID 17339554
- [Background] Mascle S, Schnell F, Thebault C, Corbineau H, Laurent M, Hamonic S, Veillard D, Mabo P, Leguerrier A, Donal E. Predictive value of global longitudinal strain in a surgical population of organic mitral regurgitation. J Am Soc Echocardiogr. 2012 Jul;25(7):766-72. doi: 10.1016/j.echo.2012.04.009. Epub 2012 May 19. PMID 22609096
- [Background] Donal E, Mascle S, Brunet A, Thebault C, Corbineau H, Laurent M, Leguerrier A, Mabo P. Prediction of left ventricular ejection fraction 6 months after surgical correction of organic mitral regurgitation: the value of exercise echocardiography and deformation imaging. Eur Heart J Cardiovasc Imaging. 2012 Nov;13(11):922-30. doi: 10.1093/ehjci/jes068. Epub 2012 Apr 14. PMID 22504944
- [Background] Magne J, Mahjoub H, Dulgheru R, Pibarot P, Pierard LA, Lancellotti P. Left ventricular contractile reserve in asymptomatic primary mitral regurgitation. Eur Heart J. 2014 Jun 21;35(24):1608-16. doi: 10.1093/eurheartj/eht345. Epub 2013 Sep 7. PMID 24014387
- [Background] Toubal O, Mahjoub H, Thebault C, Clavel MA, Dahou A, Magne J, O'Connor K, Beaudoin J, Bernier M, Le Ven F, Pibarot P. Increasing Pulmonary Arterial Pressure at Low Level of Exercise in Asymptomatic, Organic Mitral Regurgitation. J Am Coll Cardiol. 2018 Feb 13;71(6):700-701. doi: 10.1016/j.jacc.2017.11.062. No abstract available. PMID 29420967
- [Background] Clemenceau A, Berube JC, Belanger P, Gaudreault N, Lamontagne M, Toubal O, Clavel MA, Capoulade R, Mathieu P, Pibarot P, Bosse Y. Deleterious variants in DCHS1 are prevalent in sporadic cases of mitral valve prolapse. Mol Genet Genomic Med. 2018 Jan;6(1):114-120. doi: 10.1002/mgg3.347. Epub 2017 Dec 10. PMID 29224215
- [Background] Dupuis M, Mahjoub H, Clavel MA, Cote N, Toubal O, Tastet L, Dumesnil JG, O'Connor K, Dahou A, Thebault C, Belanger C, Beaudoin J, Arsenault M, Bernier M, Pibarot P. Forward Left Ventricular Ejection Fraction: A Simple Risk Marker in Patients With Primary Mitral Regurgitation. J Am Heart Assoc. 2017 Oct 27;6(11):e006309. doi: 10.1161/JAHA.117.006309. PMID 29079561